CLINICAL TRIAL: NCT05793853
Title: Advancing Product Development for Hypoparathyroidism: A Prospective Natural History Study of the Clinical Outcomes and Regulation of Disordered Mineral Metabolism
Brief Title: Hypoparathyroidism Natural History Study
Acronym: SHINE
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Mishaela Rubin, Professor of Medicine, Columbia University
Other Study IDs: AAAU3302; R01FD007629 (FDA)
Record Dates: First submitted 2022-12-23; First posted 2023-03-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypoparathyroidism Subjects: Patients who have the disease hypoparathyroidism, who are being followed to monitor various aspects of the disease over time. No interventions.
- Control Subjects: Healthy individuals to be followed to compare to hypoparathyroidism patients

SUMMARY:
This is a prospective three-year natural history study of adults with hypoparathyroidism. The goal is to monitor patients with hypoparathyroidism to define end-organ damage in the context of the disease.

The study objectives are to:

1. Build a prospective cohort of patients to study HPT-associated end-organ damage.
2. Determine end-organ physiologic consequences of HPT.
3. Elucidate determinants of HPT-associated end-organ damage.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
The goal of this study is to prospectively collect data on the natural history of hypoparathyroidism (HPT). This will enable longitudinal data collection of complications in this disease, specifically defining the epidemiology of end-organ complications of HPT that are related to high calcification propensity. It will also determine relationships between calcification burden and end-organ disease severity and progression risk and assess the utility of traditional and novel biomarkers of mineral and bone metabolism on disease diagnosis and monitoring. These data will inform future investigations on the development, study, and implementation of HPT end-organ disease modifying strategies and impact clinical practice in hypoparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability and willingness to fully comply with study procedures and restrictions.
* Ability to voluntarily provide written, signed and dated informed consent as applicable to participate in the study.
* Male or female ≥18 years of age with HPT. All HPT sub-types are eligible, including surgical (HPT-S) and nonsurgical (HPT-NS) HPT: autoimmune, genetic (including but not limited to: DiGeorge syndrome, autoimmune polyendocrine syndrome type 1, hypoparathyroidism sensorineural deafness and renal disease syndrome, Kearns-Sayre syndrome, mitochondrial encephalomyopathy with lactic acidosis and stroke-like episodes [MELAS] syndrome, mitochondrial trifunctional protein [MTP] deficiency syndrome, Kenny-Caffey syndrome, Sanjad-Sakati syndrome, autosomal dominant hypocalcemia), infiltrative (granulomatous), mineral deposition (copper, iron), metastatic, radiation and idiopathic HPT.
* Diagnosis of HPT established based on historic hypocalcemia in the setting of inappropriately low serum PTH levels on two occasions.
* All treatment regimens are permitted, including but not limited to conventional management with calcium (e.g. calcium citrate, calcium carbonate, etc), active vitamin D (calcitriol, alfacalcidol), parent vitamin D, magnesium, phosphate binders and thiazides. Use of PTH-like drugs are permitted.

Exclusion Criteria:

* Functional HPT
* Transient HPT
* Pseudohypoparathyroidism
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female ≥18 years of age with all hypoparathyroidism sub-types. Healthy male and female controls.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Kidney function | baseline, 6, 12, 18, 24, 30, 36 Months
  blood test for changes in eGFR (in mL/min/1.73m^2)

SECONDARY OUTCOMES:
Kidney calcification | Baseline and 36 Months
  Changes in kidney calcification and stones will be assessed by abdominal CT in an optional imaging sub group. Results will be assessed and reported by a clinician.
Brain calcification | Baseline and 36 Months
  Changes in brain calcification will be assessed by head CT in an optional imaging sub-group. Results will be assessed and reported by a clinician.
Vascular calcification | Baseline and 36 Months
  Changes in vascular calcification will be assessed by leg arterial calcifications on high resolution quantitative computed tomography in all, and aortic calcifications on abdominal CT and vertebral fracture assessment by DXA in optional imaging sub-group
Bone mineral density | Baseline and 36 Months
  Changes in dual energy X-ray absorptiometry will be assessed in an optional imaging sub-group
Bone microarchitecture and bone strength | Baseline and 36 Months
  Changes in high resolution peripheral quantitative computed tomography will be assessed
Cardiac function | Baseline and 36 Months
  Changes in EKG will be assessed
Transcriptomic signaling for calcification | Baseline and 36 Months
  Changes in microRNA will be assessed
Biomarkers blood | baseline, 6, 12, 18, 24, 30, 36 Months
  Changes in complete metabolic panel to see changes with eGFR (including albumin-corrected serum calcium), PTH, phosphorus, magnesium, 25(OH)D, 25(OH)D2, TSH, FT4.
Biomarkers urine | baseline, 6, 12, 18, 24, 30, 36 Months
  24 hour urine will be collected for changes in calcium, creatinine, total volume and protein
Dietary Intake | baseline, 12, 24 and 36 Months
  Food frequency questionnaires will be administered to measure changes in calcium, phosphorus, vitamin D, and sodium intake
Cognitive Function | baseline, 12, 24 and 36 Months
  Changes in cognitive function will be assessed by NIH Toolbox®; Letter Fluency by the Controlled Oral Word Association Test with the letters FAS; Sematic Fluency by Animal Fluency; List Learning and Memory by the Hopkins Verbal Learning Test; subjective cognitive function by FACT-Cog
Neurologic Tests of Motor Function | baseline, 12, 24 and 36 Months
  Repeated Chair Stand (RCS) test will be administered to see how many times a patient can sit in and stand from a chair in 30 seconds and "Timed Up and Go" Test will measure how many seconds it takes for a patient to walk to assess changes in motor function
Quality of Life Through Self-Reported Questionnaires | baseline, 12, 24 and 36 Months
  Quality of life will be assessed by SF-36, FACIT-IF (self-reported fatigue), PGI-S and PGI-I (patient global impression of severity and impact), Hospital Anxiety and Depression Scale (HADS) and the HPT Symptom Diary and changes will be tracked through visits
Calcioprotein Maturation Time | Baseline and 36 months
  Will be obtained through blood collection and measured in minutes and changes will be tracked through visits
Sclerostin | Baseline and 36 months
  Will be obtained through blood collection and measured in pmol/L and changes will be tracked through visits
FGF23 | Baseline and 36 months
  Will be obtained through blood collection and measured in pg/mL and changes will be tracked through visits

CONTACTS AND LOCATIONS:
Overall Officials: Mishaela Rubin, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center - Harkness Pavillion, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided